CLINICAL TRIAL: NCT00066781
Title: A Phase II Study Of Gemcitabine (GEMZAR) And Irinotecan (CPT-11) In Previously Untreated Patients With Measurable Disease With Unknown Primary Carcinoma
Brief Title: Gemcitabine and Irinotecan in Treating Patients With Cancer of Unknown Primary
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N004E; NCI-2011-01592 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000318830 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Carcinoma of Unknown Primary
Keywords: adenocarcinoma of unknown primary; newly diagnosed carcinoma of unknown primary; squamous cell carcinoma of unknown primary; undifferentiated carcinoma of unknown primary
MeSH Terms: conditions — Neoplasms, Unknown Primary | interventions — Gemcitabine; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort I (closed to accrual 11/17/05) (Experimental): Patients receive gemcitabine IV over 30 minutes and irinotecan IV over 90 minutes on days 1, 8, 15, and 22. Irinotecan dose may be escalated or de-escalated after course 1 depending on toxicity. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gemcitabine hydrochloride; Drug: irinotecan hydrochloride
- Cohort II (Experimental): Patients receive gemcitabine IV over 30 minutes and irinotecan IV over 90 minutes on days 1, 8, and 15. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gemcitabine hydrochloride; Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given IV
Drug: irinotecan hydrochloride — Given IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as gemcitabine and irinotecan use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with irinotecan works in treating patients with cancer of unknown primary origin.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with carcinoma of unknown primary when treated with gemcitabine and irinotecan.
* Determine the adverse event profile and tolerability of this regimen, based on the presence or absence of the UGT1A1*28 polymorphism, in these patients. (Cohort I closed to accrual 11/17/05)
* Determine the adverse event profile and tolerability of this regimen. (Cohort II)

Secondary

* Determine the time to progression and overall survival of patients treated with this regimen.
* Correlate patterns of immunohistochemical staining with response in patients treated with this regimen.
* Correlate variation in multiple different genes, whose protein products are involved in the uptake, metabolism, and distribution of these drugs, with clinical outcomes, in terms of response and toxicity, in these patients.
* Determine primary origin of cancer of unknown primary samples by completing a 92-gene RT-PCR cancer classification assay.
* Determine whether the 92-gene assay results are correlated with clinical response to gemcitabine and irinotecan.

OUTLINE:

* Cohort I (closed to accrual 11/17/05): Patients receive gemcitabine IV over 30 minutes and irinotecan IV over 90 minutes on days 1, 8, 15, and 22. Irinotecan dose may be escalated or de-escalated after course 1 depending on toxicity. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
* Cohort II: Patients receive gemcitabine IV over 30 minutes and irinotecan IV over 90 minutes on days 1, 8, and 15. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed carcinoma of undetermined origin, with any of the following light microscopic diagnoses:

  * Adenocarcinoma

    * Poorly differentiated non-small cell carcinoma
    * Poorly differentiated squamous cell carcinoma
* Primary site not revealed by the following diagnostic tests:

  * Complete history and physical
  * Complete blood count and chemistries
  * Chest x-ray and/or CT scan
  * Abdominal CT scan
  * Directed evaluation of symptomatic areas
  * Mammogram in women
  * Colonoscopy in patients with liver metastases to exclude a colon primary
  * Hematoxylin and eosin (H&E) staining OR immunostaining if H&E results are unclear, including all of the following:

    * Keratin or epithelial membrane antigen
    * S-100 or HMB45
    * LCA (CD45)
    * Chromogranin or synaptophysin
    * Thyroid transcription factor 1
* Measurable disease
* Patients with any of the following conditions are not eligible:

  * Neuroendocrine tumors
  * Women with axillary node involvement only
  * Women with adenocarcinoma of the peritoneum
  * Carcinoma involving only 1 site, with resectable tumor at that site
  * Squamous cell carcinoma limited to cervical, supraclavicular, or inguinal lymph nodes
  * Men with poorly differentiated mediastinal or retroperitoneal tumor with stains suggestive of germ cell origin or serum tumor markers (AFP/HCG)
  * Men with prominent blastic bony metastases or markedly elevated prostate-specific antigen, suggesting prostate origin
* Must be willing to provide blood and tissue samples
* No brain or meningeal involvement

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin must meet 1 of the following criteria:

  * Less than or equal to upper limit of normal (ULN) and no UGT1A1 genotyping is required
  * Greater than ULN but less than 2 times ULN and UGT1A1 for 6/7 genotype or 7/7 genotype patients
* Alkaline phosphatase no greater than 3 times ULN
* AST no greater than 3 times ULN (5 times ULN if liver metastases are present)

Renal

* Creatinine no greater than 2.0 times ULN

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other invasive malignancy within the past 5 years
* No other severe concurrent disease that would make the patient inappropriate for the study in the judgment of the investigator
* No uncontrolled infection

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent biologic agents
* No concurrent filgrastim (G-CSF)

Chemotherapy

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to more than 25% of the bone marrow
* No concurrent radiotherapy

Surgery

* More than 4 weeks since prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2004-02; Primary Completion 2008-04 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P. Goetz, MD, Study Chair — Mayo Clinic
Locations (4):
- United States (4):
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska

REFERENCES:
- [Result] Holtan SG, Foster NR, Erlichman CE, et al.: Gemcitabine (G) and irinotecan (CPT-11) as first-line therapy for carcinoma (ca) of unknown primary (CUP): An NCCTG phase II trial. [Abstract] J Clin Oncol 26 (Suppl 15): A-13525, 2008.
- [Derived] Holtan SG, Steen PD, Foster NR, Erlichman C, Medeiros F, Ames MM, Safgren SL, Graham DL, Behrens RJ, Goetz MP. Gemcitabine and irinotecan as first-line therapy for carcinoma of unknown primary: results of a multicenter phase II trial. PLoS One. 2012;7(7):e39285. doi: 10.1371/journal.pone.0039285. Epub 2012 Jul 17. PMID 22815703

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort I: Patients receive gemcitabine IV over 30 minutes and irinotecan IV over 90 minutes on days 1, 8, 15, and 22. Irinotecan dose may be escalated or de-escalated after course 1 depending on toxicity. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Cohort I | Cohort II
Started | 14 | 17
Completed | 14 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I | Cohort II | Total
Number analyzed (Participants) | 14 | 17 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (9) | 61 (15) | 62 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 8 | 9 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 13 | 15 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Response Rate (Partial or Complete Response for 2 Consecutive Evaluations at Least 4 Weeks Apart) as Measured by RECIST Criteria
Description: The primary endpoint is confirmed response rate. If measurable disease is present, a confirmed tumor response is defined to be either a CR or PR noted as the objective status on 2 consecutive evaluations at least 4 weeks apart. All registered patients meeting the eligibility criteria that have signed a consent form and have begun treatment will be evaluable for response.
Time Frame: Up to 2 years
Population: All evaluable patients
Measure: Number (95% Confidence Interval); unit: percentage of patients with response
Arm/Group | Cohort I | Cohort II
Number analyzed (Participants) | 11 | 15
percentage of patients with response | 9 [0 to 41] | 13 [2 to 40]

2. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as the time from registration to death due> to any cause. The distribution of survival time will be estimated using> the method of Kaplan-Meier . Overall survival will be calculated for> all evaluable patients combined and by group (ie. for patients with or> without the UGT1A1*28 polymorphism).
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort I | Cohort II
Number analyzed (Participants) | 11 | 15
Months | 4 [2.2 to 15.6] | 9.3 [4.1 to 12.1]

3. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression is defined as the time from registration to documentation of disease progression. If a patient dies without a documentation of disease progression, the patient will be considered to have had tumor progression at the time of their death unless there is sufficient documented evidence to conclude no progression occurred prior to death. If the patient is declared to be a major treatment violation, the patient will be censored on the date the treatment violation was declared to have occurred. In the case of a patient starting treatment and then never returning for any evaluations, the patient will be censored for progression on day 1 post-registration. The distribution of time to progression will be estimated using the method of Kaplan-Meier. Time to disease progression will be calculated for all evaluable patients combined and by group (ie. for patients with or without the UGT1A1*28 polymorphism).
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort I | Cohort II
Number analyzed (Participants) | 11 | 15
Months | 3.7 [1.7 to 7.8] | 3.4 [1.6 to 9.3]

ADVERSE EVENTS:
Arm/Group | Cohort I | Cohort II
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/17
Other Adverse Events (participants affected / at risk) | 14/14 | 16/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I (N=14) | Cohort II (N=17)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 4 (5) | 3 (3)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 5 (5)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 9 (13) | 12 (14)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (9) | 7 (8)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (7) | 8 (9)
Edema limbs (General disorders) | 0 (0) | 3 (6)
Fatigue (General disorders) | 6 (10) | 7 (14)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (1) | 2 (2)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 4 (8) | 3 (3)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (5)
Neutrophil count decreased (Investigations) | 4 (7) | 2 (2)
Platelet count decreased (Investigations) | 3 (4) | 3 (4)
Weight gain (Investigations) | 2 (3) | 2 (3)
Weight loss (Investigations) | 3 (4) | 5 (6)
Anorexia (Metabolism and nutrition disorders) | 10 (14) | 12 (19)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 6 (10) | 2 (4)
Peripheral ischemia (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes